CLINICAL TRIAL: NCT05074823
Title: Analgesic Effects of Three Different Doses of Intrathecal Ketamine as an Adjuvant to Intrathecal Bupivacaine in Patients Undergoing Knee Arthroscopy. A Randomized Prospective Double-blinded Study
Brief Title: Comparing Three Different Doses of Intrathecal Ketamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, associate professor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Ketamine 3 doses
Record Dates: First submitted 2021-09-22; First posted 2021-10-12 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Ketamine Causing Adverse Effects in Therapeutic Use
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketamine 0.1 (Active Comparator): Group I: will include 35 patients, will receive 3mL of bupivacaine (heavy) 0.5% in addition to 0.5 ml of a preservative-free ketamine 0.1 mg/kg
  Interventions: Drug: Ketamine 0.1 mg
- Ketamine 0.2 (Active Comparator): Group II will include 35 patients, will receive 3mL of bupivacaine (heavy) 0.5% in addition to 0.5 ml of a preservative-free ketamine 0.2 mg/kg
  Interventions: Drug: Ketamine 0.2 mg
- Ketamine 0.3 (Active Comparator): Group III will include 35 patients, will receive 3mL of bupivacaine (heavy) 0.5% in addition to 0.5 ml of a preservative-free ketamine 0.3 mg/kg
  Interventions: Drug: Ketamine 0.3 mg

INTERVENTIONS:
Drug: Ketamine 0.1 mg — Patients will receive 3mL of bupivacaine (heavy) 0.5% in addition to 0.5 ml of a preservative-free ketamine 0.1 mg/kg
  Arms: Ketamine 0.1
Drug: Ketamine 0.2 mg — will receive 3mL of bupivacaine (heavy) 0.5% in addition to 0.5 ml of a preservative-free ketamine 0.2 mg/kg
  Arms: Ketamine 0.2
Drug: Ketamine 0.3 mg — will receive 3mL of bupivacaine (heavy) 0.5% in addition to 0.5 ml of a preservative-free ketamine 0.3 mg/kg
  Arms: Ketamine 0.3

SUMMARY:
The aim of this study is to compare the postoperative analgesic effect of three different doses of intrathecal ketamine as an adjuvant to bupivacaine in patients undergoing knee arthroscopy.

DETAILED DESCRIPTION:
A meta-analysis of adult human randomized controlled studies that compared single dose perioperative intrathecal ketamine plus intrathecal bupivacaine to bupivacaine alone in spinal anesthesia suggests that there is a benefit to using intrathecal ketamine as an adjunct to bupivacaine in multimodal analgesia. However, there are still knowledge and experience gaps regarding neuraxial ketamine dosing in this regard.

Aim of the study:

The aim of this study is to compare the postoperative analgesic effect of three different doses of intrathecal ketamine as an adjuvant to bupivacaine in patients undergoing knee arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years.
* BMI: 20-30 kg.m2
* Sex: both males and females.
* ASA physical status: I-III.
* Operation: knee arthroscopy.

Exclusion Criteria:

* Patient's refusal to participate in the study.
* Aged less than 18 years,
* known allergy to L.A.,
* Coagulopathy or thrombocytopenia,
* height less than 150 cm, morbidly obese infection at the site of injection.
* Chronic pain syndromes,
* pregnant woman
* Patients on regular use of analgesic or who received analgesic 24 h before surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-02-26 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic request | First 24 hours
  From the time of intrathecal administration of the drug to the time of patient needs the first rescue analgesic drug

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided